CLINICAL TRIAL: NCT06007586
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study on Prevention and Treatment of CINV Induced by TC Regimen in Gynecological Malignant Tumors
Brief Title: Prevention and Treatment of CINV Caused by TC Regimen in Gynecological Malignant Tumor Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: the Norman Bethune's "Research Wing Promotion"-Supporting Research Projects (Unknown); Peking Union Medical College Hospital Talent Cultivation Program (Unknown); Medical High Level Talents Program (Unknown); Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Dengfeng Wang, Deputy chief, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CINV202306
Record Dates: First submitted 2023-08-11; First posted 2023-08-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Gynecological Tumor; Ovarian Cancer; Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer
Keywords: Gynecologic Cancer; chemotherapy-induced nausea and vomiting; Paclitaxel-carboplatin
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Vomiting | interventions — Aprepitant; Dexamethasone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both patients and investigators, including follow-up staff, were blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): patients in group A received the two-drug antiemetic regimen (placebo cycle) during the first cycle followed by the three-drug regimen (aprepitant cycle) during the second cycle.
  The two-drug regimen (placebo cycle) consisted of intravenous placebo 130 mg, intravenous ondansetron 8 mg, and intravenous dexamethasone 12 mg, all administered 30 minutes before chemotherapy on day 1, followed by oral dexamethasone 8 mg once daily on days 2-4.
  The three-drug regimen (aprepitant cycle) replaced placebo with intravenous aprepitant 130 mg on day 1, with all other medications administered as in the two-drug regime
  Interventions: Drug: Aprepitant Injection
- Group B (Experimental): patients in group B received the regimens in the reverse order. The three-drug regimen (aprepitant cycle) replaced placebo with intravenous aprepitant 130 mg on day 1, with all other medications administered as in the two-drug regime.
  The two-drug regimen (placebo cycle) consisted of intravenous placebo 130 mg, intravenous ondansetron 8 mg, and intravenous dexamethasone 12 mg, all administered 30 minutes before chemotherapy on day 1, followed by oral dexamethasone 8 mg once daily on days 2-4.
  Interventions: Drug: Aprepitant Injection

INTERVENTIONS:
Drug: Aprepitant Injection — Two antiemetic groups use placebo, dexamethasone and ondansetron. Three antiemetic groups use aprepitant, dexamethasone and ondansetron.
  Other Names: dexamethasone; ondansetron

SUMMARY:
To determine the best method to prevent CINV caused by TC regimen in patients with gynecological malignant tumor.

Paclitaxel-carboplatin (TC) is the most widely used regimen for gynecologic malignancies, yet chemotherapy-induced nausea and vomiting (CINV) remain common and distressing. Optimal prophylaxis is uncertain. This trial evaluated whether adding the NK1 receptor antagonist aprepitant to standard two-drug prophylaxis (5-HT3 receptor antagonist plus dexamethasone) improves CINV control.

DETAILED DESCRIPTION:
The risk of vomiting caused by high-dose carboplatin is controversial, and there is currently no prevention of TC in patients with gynecological malignant tumors High-level evidence-based medical evidence for programme-induced CINV. Therefore, different guidelines recommend the best antiemetic regimen as well It's different. This study is intended to conduct a prospective, multicenter, randomized, double-blind, placebo-controlled, crossover study The designed Phase III clinical study provides important data and basis for clinical practice and guideline formulation.

In this prospective, multicenter, double-blind, placebo-controlled, crossover phase III trial, patients with gynecologic malignancies scheduled for at least two cycles of TC were randomly assigned to receive aprepitant or placebo with ondansetron and dexamethasone during cycle 1, crossing over to the alternate regimen in cycle 2. The primary endpoint was complete response (CR: no emesis, no significant nausea and no rescue therapy) in the delayed phase (24-168 hours). Secondary endpoints included CR in acute and overall phases, nausea severity, rescue medication use, adverse events, and patient satisfaction.

ELIGIBILITY:
Eligibility criteria: histologically confirmed gynecologic malignancies (including newly diagnosed cases and recurrent cases without chemo- or radiotherapy within the past six months); age 20-75 years; ECOG performance status 0-2; scheduled to receive at least two cycles of paclitaxel (175 mg/m²) plus carboplatin (AUC 5-6) every 3 weeks; and adequate organ function (bilirubin and creatinine within normal range, ALT and AST < 2× upper limit of normal).

Exclusion criteria: included prior chemotherapy, radiotherapy, or targeted therapy for the current recurrence; known brain metastases or history of brain tumors; history of gastrointestinal malignancy or major gastrointestinal surgery (except polypectomy or appendectomy); incomplete bowel obstruction; vestibular dysfunction; massive ascites (unless drained); concomitant opioid use; or diabetes mellitus.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 143 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) rate in the delayed period | 24 hours to 7days after chemotherapy (each cycle is 21 days)
  CR is defined as no emesis, no significant nausea (VAS ≤4, where 0 = none, 10= = most severe), and no use of rescue antiemetics.

SECONDARY OUTCOMES:
CR rates in the acute phase (0-24 hours) and overall phase (0-7 days). | acute phase: within 24 hours after chemotherapy (each cycle is 21 days); overall phase: within 7 days after chemotherapy (each cycle is 21 days).
  CR rates in the acute phase (0-24 hours) and overall phase (0-7 days).
the use of rescue antiemetic | within 7 days after chemotherapy (each cycle is 21 days).
  the use of rescue antiemetic (0-7 days)
patient satisfaction | On day 7 and 14 of each cycle (each cycle is 21 days).
  patient satisfaction assessed with a 7-point Likert-type scale (1=Very dissatisfied; 2=dissatisfied; 3=Relatively dissatisfied; 4=quite satisfied; 5=somewhat satisfied; 6=Satisfied; 7=Very satisfied)
AEs | within 7 days after chemotherapy (each cycle is 21 days).
  incidence of adverse events
severity of nausea | within 7 days after chemotherapy (each cycle is 21 days).
  severity of nausea (VAS: 0 = none, 10 = most severe)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Dengfeng Wang, Chengdu, Sichua
  - Sichuan Cancer Hospital, Chengdu

IPD SHARING:
Plan to Share IPD: No